CLINICAL TRIAL: NCT01499134
Title: Effect of Nebivolol Compared With Metoprolol in Hypertensive Patients With Peripheral Arterial Disease
Brief Title: Comparison of 2 Beta Blocker Drugs on Peripheral Arterial Disease in Patients With High Blood Pressure
Acronym: ENCOMPASS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11C.18
Record Dates: First submitted 2011-10-24; First posted 2011-12-26 (Estimated); Results first posted 2014-12-03 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-12

CONDITIONS: Peripheral Artery Disease; Hypertension
MeSH Terms: conditions — Peripheral Arterial Disease; Hypertension | interventions — Nebivolol; Metoprolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- nebivolol (Experimental): nebivolol 1 to 4 capsules daily
  Interventions: Drug: nebivolol
- metoprolol succinate (Active Comparator): metoprolol 1 to 4 capsules daily
  Interventions: Drug: Metoprolol succinate

INTERVENTIONS:
Drug: nebivolol — Study medication will initially be dispensed as one capsule daily and the dose will be titrated at the study visits. Nebivolol is approved for hypertension treatment at a dose of 5-40 mg daily. Based on the study titration schedule, the maximum doses used will be 20 mg of nebivolol (each maximum dose being contained in 4 capsules for daily dosing).
  Other Names: Bystolic
  Arms: nebivolol
Drug: Metoprolol succinate — Study medication will initially be dispensed as one capsule daily and the dose will be titrated at study visits. Metoprolol succinate at 25-400 mg daily. Based on the study titration schedule, the maximum dose used will be 200 mg of metoprolol succinate (each maximum dose being contained in 4 capsules for daily dosing).
  Other Names: Toprol XL
  Arms: metoprolol succinate

SUMMARY:
This is a 26-week, prospective double-blind, randomized pilot trial of nebivolol versus an active control, metoprolol succinate, in patients with established lower-extremity peripheral artery disease, hypertension, and at least moderate risk for coronary artery disease.

DETAILED DESCRIPTION:
Peripheral arterial disease (PAD) affects up to an estimated 16-29% of men and women over age 50, and is associated with increased cardiovascular morbidity and mortality. Beta-blockers have been shown to reduce the risk of myocardial infarction and death in patients with coronary artery disease (CAD) and are indicated for the treatment of hypertension in patients with PAD. However, there is a theoretical risk that antihypertensive therapy may decrease limb perfusion pressure and therefore exacerbate symptoms of claudication or limb ischemia. Patients with CAD and concomitant PAD are less likely to be prescribed beta-blockers, even though most patients are able to tolerate antihypertensive therapy without worsening of symptoms.

The third generation beta-blocker, nebivolol, has vasodilating properties in addition to beta-adrenergic blockade. This vasodilatory effect is mediated through the L-arginine-nitric oxide-dependent pathway. Nitric oxide is a critical modulator of vascular disease with effects that lead to vasodilatation, endothelial regeneration, inhibition of leukocyte chemotaxis and inhibition of platelet adhesion. This combination of beta-blockade and nitric oxide-dependent vasodilation may enhance effectiveness and tolerability of nebivolol versus other beta-blockers in patients with hypertension, CAD or high-risk state, and PAD.

This study will be a pilot comparative effectiveness study to examine the effect of nebivolol versus metoprolol succinate in patients with lower-extremity PAD and at least moderate risk for CAD on PAD symptoms as measured by both functional and quality of life measures.

ELIGIBILITY:
Inclusion Criteria:

* Men and non-pregnant, non-lactating women 45 years of age or older
* Able to give informed consent and complete scheduled visits
* Mild-moderate bilateral lower extremity peripheral arterial disease as defined by an ankle-brachial index (ABI measurement of 0.6-0.9. If a subject has baseline claudication symptoms, the symptoms must be stable for the 3 months preceding enrollment.
* History of hypertension. Blood pressure at the screening visit must be ≤160/100 mmHg and ≥100/60 mmHg for all subjects. If a subject is currently prescribed beta-blocker therapy, BP at the screening visit must be ≤140/90 mmHg. In addition, heart rate must be ≥55 beats per minute if currently prescribed a beta-blocker and ≤60 beats per minute if not currently prescribed a beta-blocker.
* At least moderate risk for CAD.

Exclusion Criteria:

* Participation in another clinical trial
* Ongoing ischemic (resting) limb pain, or lower extremity ulceration due to arterial insufficiency, or an ABI indicating <0.6 indicating disease potentially requiring revascularization
* History of limb or digit amputation due to arterial insufficiency
* Revascularization of peripheral vessels within the preceding 6 months
* Uncontrolled hypertension as defined by systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg
* Contraindication or allergy to beta blocker therapy
* History of myocardial infarction , coronary revascularization, or a cerebrovascular event within the preceding 6 months
* Class III or IV angina
* Current or past history of New York Heart Association (NYHA) class III or IV heart failure
* Inability to walk on a treadmill for any reason
* Regular use of nitroglycerin or nitrates including oral, transdermal ointment or patch, or sublingual, translingual spray and/or combination agents containing nitrates
* Active liver, pulmonary, infectious or inflammatory process
* History of malignancy within preceding 5 years (excluding basal or squamous cell skin cancer)
* History of any other condition that, in the opinion of the investigators, renders it unsafe for the subject to be enrolled

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2011-08; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Duffy, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nebivolol | Metoprolol Succinate
Started | 9 | 8
Completed | 9 | 7
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Original sample size for pilot study was fixed at 40 subjects. Lagging enrollment necessitated completion at 17 subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nebivolol | Metoprolol Succinate | Total
Number analyzed (Participants) | 9 | 8 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (8) | 65 (8) | 66 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 2 | 9
  Male | 2 | 6 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 8 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 3 | 8
  White | 4 | 5 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 8 | 17

OUTCOME MEASURES:

1. Primary Outcome: Peak Walking Time (PWT)
Description: Change in peak walking time (PWT) is measured in seconds. The PWT is defined as when walking on a treadmill cannot continue due to maximal leg pain, resulting in the discontinuation of the treadmill test.
Time Frame: Baseline PWT is measured at the time of enrollment and again at the final study visit at 26 weeks.
Population: One patient in the metoprolol succinate group withdrew consent prior to the end of the study, therefore, only 7 participants are included in the analysis for this group.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Nebivolol | Metoprolol Succinate
Number analyzed (Participants) | 9 | 7
seconds | 110.4 (89.7) | -19.4 (110.8)
Statistical Analysis 1: Comparison: Nebivolol vs Metoprolol Succinate; Test type: Superiority or Other; p = 0.039, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Ankle-brachial Index (ABI)
Description: Change in measurement of Ankle-brachial index (ABI). The ABI is the ratio of the blood pressure measured in the lower legs to the blood pressure measured in the arms.
Time Frame: Baseline ABI is measured at the time of enrollment and again at the final study visit at 26 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ankle-Brachial Index
Arm/Group | Nebivolol | Metoprolol Succinate
Number analyzed (Participants) | 9 | 7
Ankle-Brachial Index | 0.03 (0.14) | 0.06 (0.11)
Statistical Analysis 1: Comparison: Nebivolol vs Metoprolol Succinate; Test type: Superiority or Other; p = 0.585, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Claudication Onset Time (COT)
Description: Change in measurement of claudication onset time (COT). The COT is defined as the time when a patient first experienced pain walking during a treadmill test.
Time Frame: Baseline COT is measured at the time of enrollment and again at the final study visit at 26 weeks.
Population: Final measurements of COT in the metoprolol succinate group excludes one subject who did not experience claudication while walking during the treadmill test, and one subject who withdrew consent prior to the end of the study, therefore, only 6 participants are included in the analysis for this group.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Nebivolol | Metoprolol Succinate
Number analyzed (Participants) | 9 | 6
seconds | 155.7 (217.5) | 148.7 (173.1)
Statistical Analysis 1: Comparison: Nebivolol vs Metoprolol Succinate; Test type: Superiority or Other; p = 1.000, Wilcoxon (Mann-Whitney) — This p-value is correct, confirmed with report from statistician

4. Secondary Outcome: Walking Impairment Questionnaire (WIQ) - Change Calf Pain
Description: Change in calf pain as captured by the Walking Impairment Questionnaire (WIQ). A 5 point Likert scale scoring ranges from 1) No Difficulty, 2) Slight Difficulty, 3) Some Difficulty, 4) Much Difficulty, and 5) Great Difficulty. The scores are determined by dividing the score by the maximum possible score and then multiplying by 100. The score ranges from 0-100 with lower scores indicating greater pain.
Time Frame: Baseline WIQ is completed at the time of enrollment and again at the final study visit at 26 weeks.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nebivolol | Metoprolol Succinate
Number analyzed (Participants) | 9 | 7
units on a scale | 25 (28) | 10.7 (40.5)
Statistical Analysis 1: Comparison: Nebivolol vs Metoprolol Succinate; Test type: Superiority or Other; p = 0.363, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Walking Impairment Questionnaire (WIQ) - Change in Buttock Pain
Description: Change in buttock pain as captured by the Walking Impairment Questionnaire (WIQ). A 5 point Likert scale scoring ranges from 1) No Difficulty, 2) Slight Difficulty, 3) Some Difficulty, 4) Much Difficulty, and 5) Great Difficulty. The scores are determined by dividing the score by the maximum possible score and then multiplying by 100. The score ranges from 0-100 with lower scores indicating greater pain.
Time Frame: Baseline WIQ is completed at the time of enrollment and again at the final study visit at 26 weeks.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nebivolol | Metoprolol Succinate
Number analyzed (Participants) | 9 | 7
units on a scale | -8.3 (12.5) | 14.3 (19.7)
Statistical Analysis 1: Comparison: Nebivolol vs Metoprolol Succinate; Test type: Superiority or Other; p = 0.017, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Walking Impairment Questionnaire (WIQ) - Change in WIQ Distance Score
Description: Change in distance score as captured by the Walking Impairment Questionnaire (WIQ) distance score subscale. The degree of difficulty in the walking of specific distances is ranked on a 0 to 4 Likert scale, in which 0 represents the inability to walk the distance and 4 represents no difficulty. A Likert scale is an ordinal scale of consecutive, equidistant, numerical values (ie, 0 to 4). The distances assessed in the WIQ range from walking indoors around the home to walking 5 blocks (1500 feet). The items on the subscale are weighted according to the difficulty of walking. The distance score is determined by dividing the total weighted score by the greatest possible weighted score and multiplying by 100. Scores range from 0-100.
Time Frame: Baseline WIQ is completed at the time of enrollment and again at the final study visit at 26 weeks.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nebivolol | Metoprolol Succinate
Number analyzed (Participants) | 9 | 5
units on a scale | 13.52 (27.37) | 28.28 (31.18)
Statistical Analysis 1: Comparison: Nebivolol vs Metoprolol Succinate; Test type: Superiority or Other; p = 0.476, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Walking Impairment Questionnaire (WIQ) - Change in WIQ Speed Score
Description: Change in speed score as captured by the Walking Impairment Questionnaire (WIQ) speed score subscale. In the walking speed component, the degree of difficulty walking is ranked on a 0 to 4 scale where speed is assessed for each of the following speeds: at the following speeds: 1, slowly; 2, average speed; 3, quickly; or 4, running or jogging 1 block. Zero represents the inability to walk the specified speed, and 4 represents no difficulty. The items on the subscale are weighted according to the difficulty of the task. The speed score is determined by dividing the total weighted score by the greatest possible weighted score and multiplying by 100. Scores range from 0-100.
Time Frame: Baseline WIQ is completed at the time of enrollment and again at the final study visit at 26 weeks.
Population: One patient in the metoprolol succinate group withdrew consent prior to the end of the study, therefore, only 7 participants are included in the analysis for this group. One patient in the nebivolol group failed to complete the items in the WIQ speed score subscale, therefore, only 8 patients were included in the analysis for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nebivolol | Metoprolol Succinate
Number analyzed (Participants) | 8 | 7
units on a scale | 21.88 (30.08) | -6.83 (35.34)
Statistical Analysis 1: Comparison: Nebivolol vs Metoprolol Succinate; Test type: Superiority or Other; p = 0.170, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Walking Impairment Questionnaire (WIQ) - Change in WIQ Stairs Score
Description: Change in stairs score as captured by the Walking Impairment Questionnaire (WIQ) stairs subscale. This scale item asks the subject to describe the degree of difficulty climbing one, two, or three flights of stairs in the past week. A flight of stairs is defined as 14 steps. A 5 point Likert scale scoring ranges from 1) No Difficulty, 2) Slight Difficulty, 3) Some Difficulty, 4) Much Difficulty, 5) Unable to Do, or 6) Didn Do for Other Reasons. The items on the subscale are weighted according to the difficulty of the task. The stairs score is determined by dividing the total weighted score by the greatest possible weighted score and multiplying by 100. Scores range from 0-100.
Time Frame: Baseline WIQ is completed at the time of enrollment and again at the final study visit at 26 weeks.
Population: Four people in the nebivolol group and 1 person in the metoprolol group did not complete the items in the "Stairs" WIQ subscale therefore they were excluded from the analysis. One person in the metoprolol succinate group withdrew consent before the end of the study so they were also excluded from the final analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nebivolol | Metoprolol Succinate
Number analyzed (Participants) | 5 | 6
units on a scale | 21.67 (37.20) | 24.31 (38.77)
Statistical Analysis 1: Comparison: Nebivolol vs Metoprolol Succinate; Test type: Superiority or Other; p = 0.595, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Nebivolol | Metoprolol Succinate
Serious Adverse Events (participants affected / at risk) | 2/9 | 0/8
Other Adverse Events (participants affected / at risk) | 0/9 | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nebivolol (N=9) | Metoprolol Succinate (N=8)
Decrease in hemoglobin (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — The patient had a decrease in hemoglobin and was sent to outside hospital where upper endoscopy and colonoscopy found no bleeding. The patient received 2 units of packed red blood cells started on a regimen of ferrous sulfate 320 mg PO BID.
Peripheral stent placed (Vascular disorders) | 1 (1) | 0 (0) — The patient had elective left femoral and popliteal artery angioplasty with stent placed in left leg due to disabling claudication.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No